CLINICAL TRIAL: NCT07059650
Title: A Phase Ib/II, Multicenter Study to Evaluate the Efficacy and Safety of DZD8586 Combination Therapy in Diffuse Large B-cell Lymphoma
Brief Title: DZD8586 Combination Therapy in Patients With Diffuse Large B-cell Lymphoma (TAI-SHAN12)
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Dizal Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: DZ2024B0001
Record Dates: First submitted 2025-06-16; First posted 2025-07-11 (Actual); Last update posted 2025-08-28 (Actual); Status verified 2025-06

CONDITIONS: Diffuse Large B-Cell Lymphoma
MeSH Terms: conditions — Lymphoma, Large B-Cell, Diffuse

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- DZD8586 combination therapy (Experimental): 3 cohorts are included in this arm:
  Cohort 1: Treatment naïve DLBCL patients will receive DZD8586 at the protocol defined dose level, combined with R-CHOP (rituximab, cyclophosphamide, doxorubicin, vincristine, and prednisone) regimens for 6 cycles, and then DZD8586 as maintenance therapy for patients who achieved (complete response) CR or (partial response) PR after 6 cycles combination therapy.
  Cohort 2: Relapsed/refractory DLBCL patients will receive DZD8586 at the protocol defined dose level, combined with R-GemOx (rituximab, gemcitabine, and oxaliplatin) regimens for 8 cycles, and then DZD8586 as maintenance therapy for patients who achieved CR or PR after 8 cycles combination therapy.
  Cohort 3: Relapsed/refractory DLBCL patients will receive DZD8586 at the protocol defined dose level, combined with BR (bendamustine and rituximab) regimens for 6 cycles, and then DZD8586 as maintenance therapy for patients who achieved CR or PR after 6 cycles combination therapy.
  Interventions: Drug: DZD8586+R-CHOP; Drug: DZD8586+R-GemOx; Drug: DZD8586+BR

INTERVENTIONS:
Drug: DZD8586+R-CHOP — DZD8586 at the protocol defined dose level (50 mg or 75 mg, po, qd) with R-CHOP (Rituximab: 375 mg/m2, IV, d1; Cyclophosphamide: 750 mg/m2, IV, d1; Doxorubicin: 50 mg/m2, IV, d1; Vincristine: 1.4 mg/m2, IV, d1; Prednisone: 100 mg, po, d1-5) in a 21-day cycle for 6 cycles. DZD8586 (pre-defined dose level, po, qd) as maintenance therapy for CR/PR patients.
Drug: DZD8586+R-GemOx — DZD8586 at the protocol defined dose level (50 mg or 75 mg, po, qd) with R-GemOx (Rituximab: 375 mg/m2, IV, d1; Gemcitabine: 1000 mg/m2, IV, d1; Oxaliplatin: 100 mg/m2, IV, d1) in a 21-day cycle for 8 cycles. DZD8586 (pre-defined dose level, po, qd) as maintenance therapy for CR/PR patients.
Drug: DZD8586+BR — DZD8586 at the protocol defined dose level (50 mg or 75 mg, po, qd) with BR (Bendamustine: 90 mg/m2, IV, d1-d2; Rituximab: 375 mg/m2, IV, d1) in a 21-day cycle for 6 cycles. DZD8586 (pre-defined dose level, po, qd) as maintenance therapy for CR/PR patients.

SUMMARY:
This study will treat patients with diffuse large B-cell lymphoma (DLBCL). It will assess the anti-tumor efficacy and safety of DZD8586 combination therapy by using objective response rate and the incidence and severity of adverse events. It will also measure the levels of DZD8586 in the body when combined with immunochemotherapy regimens.

ELIGIBILITY:
Inclusion Criteria:

* Cohort 1:

  1. Patients with pathologically confirmed DLBCL who have not received prior anti-lymphoma therapy.
  2. Disease stage II to IV by Ann Arbor Classification.
  3. Life expectancy ≥ 12 months.
* Cohort 2, 3:

  1. Pathologically confirmed DLBCL patients who have received adequate first-line treatment containing CD20 monoclonal antibody and anthracyclines (such as R-CHOP-like regimen).
  2. Relapsed or refractory to first-line R-CHOP-like regimen.
  3. For patients who have received only one line of therapy, if the patient has not received autologous stem cell transplantation, the investigator needs to assess as unsuitable or the patient refuses intensive chemotherapy and hematopoietic stem cell transplantation.
  4. Life expectancy ≥ 6 months.
* Patients must also meet all of the following criteria to be included in this study:

  1. All patients must provide a signed and dated written informed consent prior to any study-specific procedure, sampling, and analysis.
  2. Patients must be ≥ 18 years of age at the time of informed consent.
  3. ECOG status score of 0 to 2.
  4. Presence of at least one radiologically measurable lesion in 2 perpendicular directions as assessed by CT or MRI and a positive lesion on PET/CT scan consistent with a tumor site identified by CT or MRI.
  5. Adequate bone marrow hematopoietic reserve and organ function.
  6. No uncontrolled medical complications.
  7. Patients should be able to follow the relevant requirements of this study for medication and follow-up.
  8. Willing to comply with contraceptive restrictions.

Exclusion Criteria:

* Cohort 2, 3:

  a. Hematopoietic stem cell transplantation, cell therapy, or gene therapy within 90 days prior to first dose. Radiation therapy within 14 days prior to first dose. Chemotherapy and small-molecule targeted therapy were not terminated within 5 half-lives before the first dose; macromolecule drug therapy (such as antibody therapy) was not terminated within 28 days before the first dose.
* All patients should not be included in this study if they have any of the following conditions:

  1. Indolent lymphoma-transformed DLBCL, primary mediastinal lymphoma, lymphoma involving the central nervous system, or DLBCL with MYC and BCL2 rearrangements.
  2. Prior use of BTK inhibitors.
  3. Vaccination with live attenuated vaccines or viral vector vaccines within 4 weeks prior to enrollment.
  4. Currently taking vitamin K antagonists, taking 2 or more antiplatelet/anticoagulant drugs at the same time, drugs/herbs or supplements known to potently induce or inhibit CYP3A enzyme activity, proton pump inhibitor drugs, anti-tumor traditional Chinese medicine or failing to meet the protocol-specified withdrawal time before administration in this study.
  5. Major surgery within 4 weeks or anticipated surgery after the start of this study. Or insufficiently recovered from any toxicity and/or complications of previous intervention.
  6. Clinically significant cardiac disorders. History of thrombotic diseases, stroke or intracranial hemorrhage within 6 months.
  7. Active infectious diseases.
  8. Intractable nausea and vomiting that cannot be well controlled by supportive treatment, chronic gastrointestinal diseases, dysphagia, or previous surgical resection of the intestinal segment may affect the adequate absorption of the drug.
  9. The patient has been diagnosed with other malignant diseases other than B-cell lymphoma within the past 2 years.
  10. Patients with hypersensitivity to DZD8586 drug excipients or other chemical analogues.
  11. Patients with severe or uncontrolled systemic diseases, including poorly controlled hypertension and active bleeding constitution.
  12. Serious medical or psychiatric illness that could affect participation in the study or could compromise the ability to consent
  13. Women who are pregnant or breastfeeding.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2025-08-19 (Actual); Primary Completion 2030-10 (Estimated); Study Completion 2030-10 (Estimated)

PRIMARY OUTCOMES:
Part A: Incidence and severity of adverse events | Approximately 5 years
Part B: Objective response rate (ORR) | Approximately 5 years

SECONDARY OUTCOMES:
Part A: Objective response rate (ORR) | Approximately 5 years
Part A: Complete response rate (CRR) | Approximately 5 years
Part A: Time to response (TTR) | Approximately 5 years
Part A: Duration of Response (DoR) | Approximately 5 years
Part A: Progression-Free Survival (PFS) | Approximately 5 years
Part A: Overall Survival (OS) | Approximately 5 years
Part B: Incidence and severity of adverse events | Approximately 5 years
Part B: Complete response rate (CRR) | Approximately 5 years
Part B: Time to response (TTR) | Approximately 5 years
Part B: Duration of Response (DoR) | Approximately 5 years
Part B: Progression-Free Survival (PFS) | Approximately 5 years
Part B: Overall Survival (OS) | Approximately 5 years
Part A: Peak plasma concentration (Cmax) of DZD8586 and metabolite (DZ4581) | Up to 24 hours post dose
Part A: Area under the plasma concentration versus time curve (AUC) of DZD8586 and metabolite (DZ4581) | Up to 24 hours post dose
Part A: Time to peak concentration (Tmax) of DZD8586 and metabolite (DZ4581) | Up to 24 hours post dose
Part A: Metabolite (DZ4581) to parent (DZD8586) ratio based on area under the plasma concentration versus time curve (MRAUC) | Up to 24 hours post dose
Part A: Trough concentration at steady state (Css, min) of DZD8586 and metabolite (DZ4581) | Up to 24 hours post dose
Part A: Apparent clearance at steady state (CLss/F) of DZD8586 | Up to 24 hours post dose
Part A: Accumulation index in area under the plasma concentration versus time curve (RACAUC) of DZD8586 and metabolite (DZ4581) | Up to 24 hours post dose
Part A: Accumulation index in peak plasma concentration (RACCmax) of DZD8586 and metabolite (DZ4581) | Up to 24 hours post dose

CONTACTS AND LOCATIONS:
Overall Officials: Huang, Principal Investigator — Sun Yat-sen University
Locations (16):
- China (16):
  - Peking University Third Hospital, Beijing
  - Hunan Cancer Hospital, Changsha
  - West China Hospital of Sichuan University, Chengdu
  - Chongqing Cancer Hospital, Chongqing
  - Guangdong Provincial People's Hospital, Guangzhou
  - Sun Yat-sen University Cancer Center, Guangzhou
  - Zhujiang Hospital of Southern Medical University, Guangzhou
  - The Second Affiliated Hospital Zhejiang University School of Medicine, Hangzhou
  - Anhui Provincial Cancer Hospital, Hefei
  - Shandong Cancer Hospital & Institute, Jinan
  - Linyi Cancer Hospital, Linyi
  - Shengjing Hospital of China Medical University, Shenyang
  - Shanxi Cancer Hospital, Taiyuan
  - Union Hospital, Tongji Medical College, Huazhong University of Science and Technology, Wuhan
  - The First Affiliated Hospital of Xi'an Jiaotong University, Xi'an
  - Henan Cancer Hospital, Zhengzhou

IPD SHARING:
Plan to Share IPD: No